CLINICAL TRIAL: NCT01659190
Title: The Painful Real-life Experience of the Child of Less Than Three Years During the Removal of the Collecting Bags in the Pediatric Urgency: What Strategy of Coverage?
Acronym: LINIPOCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I10028
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2012-06

CONDITIONS: Urinary Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oiled-limestone liniment (Experimental): the removal of the collecting bag is made with the Oiled-limestone liniment.
  Interventions: Other: Oiled-limestone liniment
- without Oiled-limestone liniment (No Intervention): the removal of the collecting bag is made without any special precautions

INTERVENTIONS:
Other: Oiled-limestone liniment
  Arms: Oiled-limestone liniment

SUMMARY:
Urinary infection is one of the most common bacterial infections in pediatrics and requires urine collections to be diagnosed. In France, among children under 3, urine samples are collected thanks to collecting bags.

Work teams have set as their main goal to compare the different levels of acute pain involved for children under 3 during the removing of the collecting bag, depending on the use, or not, of the Oiled-limestone liniment (randomized into 2 parallel groups), with, as a main endpoint, the difference between the results assigned to the acute pain by a pain evaluation scale (FLACC: Face-Legs-Activity-Cry-Consolability).

DETAILED DESCRIPTION:
Urinary infection is one of the most common bacterial infections in pediatrics and requires urine collections to be diagnosed. In France, among children under 3, urine samples are collected thanks to collecting bags. This nursing care, extensively recommended for young children, was the subject of a study (still in progress) in 2009 conducted by the nurses of the CHU of Limoges and the CHI of Poissy. The results have shown that the removal of the collecting bags could involve pains as severe, or even worse, as the ones observed during a urinary catheter.

The lack of documentation and stunning results of our 2009 study persuaded healthcare teams to carry on their researches and posed the following problem: the removal of the collecting bags can cause an acute pain which could result in a major discomfort for a child under 3.

In practice, the removal of the collecting bag is made without any special precautions, or with the use of several products such as the Oiled-limestone liniment. This non-medicated product, commonly used for the care of the infant seat, intra and extra hospital field, would facilitate the removal of adhesives and plasters, according to the empirical experience of caregivers. Work teams have set as their main goal to compare the different levels of acute pain involved for children under 3 during the removing of the collecting bag, depending on the use, or not, of the Oiled-limestone liniment (randomized into 2 parallel groups), with, as a main endpoint, the difference between the results assigned to the acute pain by a pain evaluation scale (FLACC: Face-Legs-Activity-Cry-Consolability).

Thanks to studies in usual care among different medical centers, that would be randomized and blindly conducted, healthcare teams would like to verify the hypothesis that the use of Oiled-limestone liniment could reduce acute pain involved in the removal of urine collecting bags among children under 36 months old. The study will be submitted to the parents of children aged 0 to 36 months old admitted to the pediatric emergency and needing a urine sample using a collecting bag.

The method of pain evaluation with the FLACC scale will be carried out as following: a caregiver will remove the collecting bag, with or without the use of the Oiled-limestone liniment, according to a prior randomized draw, and, at the same time, a second caregiver will film the care in order to provide experts assigned to measure objectively the level of the pain felt by the child during the care with videos.

Based on 136 children, during 24 months, this study would imply 3 inclusions in every medical center each month. Each inclusion should last 30 minutes.

Expected benefits would be, at first, improvement in the quality of healthcare for young children and improvement in the practice of the nurses, the nursery nurses, the auxiliaries of child welfare and the caregivers. This study would also suggests new recommendations for a good practice of nursing care, with accurate guidelines helping with the removal of collecting bags among children under 3.

ELIGIBILITY:
Inclusion Criteria:

* The children of zero in 36 months
* Children whose legal representatives accept the participation in the study
* the children must be affiliated or benefit from a health insurance scheme

Exclusion Criteria:

* Child of more than three years old
* Premature Child
* History of collection bag
* Irritated Siege
* Diarrhea

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The level of pain measured by the FLACC scale | 5 minutes

SECONDARY OUTCOMES:
Comparison at the girls and the boys of the score of the FLACC scale | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Charles LAMY, Study Director — University Hospital, Limoges
Locations (1):
- Limoges university hospital center, Limoges, France

REFERENCES:
- [Result] Lamy C, Loizeau V, Couquet C, Sturtzer C, Fluteau C, Dugas M, Labrunie A, Marin B, Desfougeres JL, Bahans C, Guigonis V, Beloni P. Pain experienced by infants and toddlers at urine collection bag removal: A randomized, controlled, clinical trial. Int J Nurs Stud. 2019 Jul;95:1-6. doi: 10.1016/j.ijnurstu.2019.03.014. Epub 2019 Mar 23. PMID 30981953